CLINICAL TRIAL: NCT00160043
Title: Phase II Open-label Study to Investigate the Efficacy and Safety of PTK787/ZK 222584 Orally Administered Once Daily or Twice Daily at 1250 mg as Second-line Monotherapy in Patients With Stage IIIB or Stage IV Non-small-cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy Study of a New Chemotherapy Agent to Treat Non Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91411; 2004-002290-22 (EudraCT Number); 308801 (Other: Company internal)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: SH T00268C
- Arm 2 (Experimental)
  Interventions: Drug: PTK787/ ZK 222584

INTERVENTIONS:
Drug: SH T00268C — 1250 mg experimental drug od
  Arms: Arm 1
Drug: PTK787/ ZK 222584 — 1250 mg experimental drug bid (500mg + 750mg)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether the study drug is effective and safe in the treatment of patients with non small cell lung cancer who have already received one platinum based chemotherapy.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer, Stage IIIB or Stage IV
* One and only 1 prior platinum-based chemotherapy
* No other uncontrolled concurrent illness
* Use of highly effective birth control methods in males or females with reproductive potential

Exclusion Criteria:

* Previous participation in another trial within the last 4 weeks
* Surgery within 10 days prior to the start of study treatment
* Brain metastases
* Confirmed diagnosis of infection with the human immunodeficiency virus (HIV)
* Current treatment with warfarin sodium (Coumadin) or similar anticoagulation medication
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (complete or partial response according to RECIST). | At baseline and every 8 weeks afterwards

SECONDARY OUTCOMES:
Time to disease progression. | At baseline and every 8 weeks afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- France (2):
  - Paris
  - Villejuif
- Germany (3):
  - Göttingen, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate

REFERENCES:
- [Result] Gauler TC, Besse B, Mauguen A, Meric JB, Gounant V, Fischer B, Overbeck TR, Krissel H, Laurent D, Tiainen M, Commo F, Soria JC, Eberhardt WEE. Phase II trial of PTK787/ZK 222584 (vatalanib) administered orally once-daily or in two divided daily doses as second-line monotherapy in relapsed or progressing patients with stage IIIB/IV non-small-cell lung cancer (NSCLC). Ann Oncol. 2012 Mar;23(3):678-687. doi: 10.1093/annonc/mdr255. Epub 2011 May 26. PMID 21617019